CLINICAL TRIAL: NCT03644628
Title: Laparoscopic Lateral Suspension Versus Laparoscopic Sacral Colpopexy for Anterior and Apical Prolapse: an International Multicentric Randomized Trial
Brief Title: Lateral Suspension Versus Sacral Colpopexy POP
Acronym: LLS vs SCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nikolaus Veit-Rubin, Senior resident Urogynecology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLS RCT 08/18
Record Dates: First submitted 2018-08-03; First posted 2018-08-23 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacropexy group (SCP) (Active Comparator): Anterior and apical repair with laparoscopic sacropexy
  Interventions: Procedure: Laparoscopic repair of anterior and apical pelvic organ prolapse
- Lateral suspension group (LLS) (Experimental): Anterior and apical repair with laparoscopic lateral suspension
  Interventions: Procedure: Laparoscopic repair of anterior and apical pelvic organ prolapse

INTERVENTIONS:
Procedure: Laparoscopic repair of anterior and apical pelvic organ prolapse — Surgical correction of anterior and apical pelvic organ prolapse by laparoscopy

SUMMARY:
The aim of the study will be to compare the SCP and LLS in the management of apical prolapse at 6 weeks, 6 months, 1 year and yearly up to 2 years with the null hypothesis being that no significant differences existed between the two surgical procedures.

DETAILED DESCRIPTION:
Background:

Pelvic Organ Prolapse (POP) is a frequent condition and can substantially affect a woman's quality of life. It is widely accepted that POP when defined by symptoms has a prevalence of 3-6 % and up to 50 % when based upon vaginal examination. Only 10 to 20 percent of affected women though seek evaluation for their condition. Although surgery is generally reserved for patients with bothersome prolapse symptoms at an advanced stage after failure of conservative treatments, a woman's lifetime risk of surgery for POP is 12-19%. Given the increasing resources that will be required for POP surgery in the future it is crucial to seek durable, cost effective interventions with minimal morbidity. Various surgical techniques exist for the correction of POP for all three compartments and there is an ongoing debate about whether to favour traditional vaginal techniques or abdominal approaches (either by laparoscopy, robotically-assisted laparoscopy or laparotomy) using synthetic mesh. Despite the 2011 FDA warning concerning POP repair with surgical mesh, transabdominal mesh procedures have not come under severe scrutiny because of more favourable risk-benefit profile. That is why sacrocolpopexy (SCP) is now considered as gold standard for the correction of apical POP and can safely and efficiently be performed laparoscopically or with robotic assistance, subsequently reducing length of hospitalization and recovery time. This technique however requires dissection at the level of the promontory, which can be challenging, particularly in obese women and when anatomical variation exists. Serious neurological or ureteral morbidity as well as life-threatening vascular injury could be the consequence of potential lesions in the sacral area. Moreover, significant dorso-lumbar pain in up to 50% of patients has been described following the use of sutures or tackers at the sacrum and most significantly, up to 30% of patients will suffer from de novo constipation due to injury to the hypogastric nerve during peritoneal dissection. Laparoscopic lateral suspension with mesh (LLS) could represent an alternative procedure, avoiding dissection at the promontory. Previous studies have shown that LLS is comparable in terms of subjective and objective outcome and that women are highly satisfied. Both procedures remain untested against each other under the rigors of a randomized controlled trial.

Hypothesis and primary objective :

The aim of the study will be to compare the SCP and LLS in the management of apical prolapse at 6 weeks, 6 months, 1 year and yearly up to 2 years with the null hypothesis being that no significant differences existed between the two surgical procedures.

Primary and secondary endpoints:

Primary outcome measures will be subjective cure of prolapse ("absence or presence of a bulge in the vagina"), objective success with anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total.

Secondary outcome measures include all other parameters such as perioperative outcomes, patient satisfaction, quality of life outcomes, complications, scores on questionnaires and reoperations.

The study protocol will be submitted to the institutional review boards of every participating study site and written informed consent will be obtained from all participants on enrolment.

Project design The investigators will perform an international multicentre single-blind randomized controlled trial with participating tertiary referral hospital centres in Italy, France, Germany and Switzerland.

PROJECT POPULATION AND STUDY PROCEDURES:

Project population, inclusion and exclusion criteria From September 2018, consecutive women referred to one of the participating centers with symptomatic stage 2 or greater apical prolapse (uterovaginal or vault prolapse) with or without anterior compartment prolapse and without significant posterior compartment prolapse will be eligible for inclusion. Exclusion criteria include those younger than 18 years of age, inability to comprehend questionnaires, to give informed consent or to return for review, unable to undergo general anesthesia, prior laparoscopic prolapse repair or vaginal mesh prolapse procedure or vaginal length less than 6 cm.

Recruitment, screening and informed consent procedure The investigators aim to end recruitment in 2020. Patients will be approached and offered participation in our study. From women who will be accepting to participate, informed consent will be obtained. Before surgery women will be examined (POP-Q) by consultant and fellows in Urogynaecology, will complete patient administered validated questionnaires. For Prolapse-related quality of life, the investigators will use the Pelvic Organ Prolapse quality of life (P-QoL) which was validated in French, Italian and German. For the assessment of lower urinary tract symptoms, the investigators will use the International consultation on incontinence questionnaire for female lower urinary tract symptoms (ICIQ-FLUTS) which was validated in French, Italian and German. For the assessment of sexual function, the investigators will use either the Female Sexual Function Index (FSFI) or the IUGA-revised Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, depending on the availability in the local language of the investigation site. The FSFI is available in French and Italian and the PISQ-IR in French and German. For the assessment of bowel dysfunction, the Wexner score will be used. All patients will undergo multichannel urodynamics including at least a free-flow study, cystometry with bladder filling to maximum of 500 mL, a stress-test in a sitting and standing position with and without prolapse reduction and a pressure-flow. Prolapse will be reduced using sponge-holding forceps at the apex. Women without symptoms of urinary stress incontinence (USI) and with positive stress test with or without prolapse reduction will be considered as having occult stress urinary in- continence (SUI). Those who will be eligible and agree to participation will complete written consent forms and will be enrolled. After completion of study consent, allocation to the SCP group or the LLS group will be done by computer generated randomization by the study statistician. The prolapse repair (SCP or LLS) will be performed either with traditional laparoscopy or with robotic assisted laparoscopy.

Clinical assessment and data collection:

Preoperative parameters will be defined as follows: Body Mass Index, Parity, Vaginal deliveries, sexual activity, dyspareunia, hormonal status, previous operations including POP surgery, hysterectomy, stress urinary incontinence, lower urinary tract symptoms such as urgency, increased daytime frequency and nycturia. Perioperative parameters will be defined as follows: operating time from knife to skin to cessation of cystoscopy. Intra- operative blood loss will be defined in milliliters by the anesthetist. All patients will have the indwelling catheter removed on day 1 and will complete a 24-hour trial of void. Patients will be discharged after a successful trial of void or successful teaching of clean intermittent self-catheterization (CISC) and not requiring analgetic injection in the last 12 hours. Catheters days will be defined as days indwelling catheter or CISC was used. Admission days will equal number of nights in hospital at midnight. Pain score at 1 month will be recorded on a visual analogue scale of 0-10 (0 no pain; 10 worst pain).

Postoperative follow-up visits will be planned at 6 weeks, 6 months, 1 year and then yearly up to 2 years.

The 6-week examination and review will be performed by the surgeon with all study data and future visits completed by blinded co-authors (Different surgeon or Urogynaecology fellows) who will be unaware of group allocation. Return to activities of daily living will be defined as days to return to driving, preparing meals, and shopping.

Women with problems will be referred by the reviewers to our clinics for management.

Self-assessed patient satisfaction (circle a score that describes your satisfaction with surgery) will be completed on a visual analogue scale (VAS) of 0-10 with 0 being lowest as previously described and using the Patient Global Impression of Improvement (PGI-I).

At every subsequent follow-up visit, patients will be interviewed about prolapse symptoms, asked to fill-out the previously mentioned questionnaires, the VAS, the PGI-I and the following parameters will be assessed: sexual activity, dyspareunia, hormonal status, operations for SUI, recurrent or de novo SUI, lower urinary tract symptoms such as urgency, increased daytime frequency and nocturia. The investigators will also report complication rates using the Clavien Dindo scale.

The investigators will follow the recommendations of the International Urogynaecology Association (IUGA) for reporting outcome of surgical procedures for pelvic organ prolapse and mesh-related complications will be classified using the joint International Urogynaecology Association/International Continence Society (IUGA/ICS) complication classification calculator.

STATISTICS AND METHODOLOGY:

Power calculation:

Given a 76% 2-year objective success rate for SP and 89% with LS, the sample size required to detect a 30% difference in success rates with a power of 80% and alpha .05 was 47 per group. To allow for drop of 15% and to ensure an adequately powered study 110 will be recruited. The study will be registered at the clinical trials registry www.clinicaltrials.gov after the enrollment of patients had commenced.

Methodology:

Frequency and percentages will be used to describe categorical variables, Fisher's exact test will be used to compare treatment groups, and logistic regression to estimate odds ratios (ORs) and associated 95% confidence intervals (95% CIs). Matched analyses for pre- and post-consistency will use McNemar test. Means and standard deviations (SDs) will be used to describe approximately normally distributed continuous data. Analysis of covariance (ANCOVA) will be used to compare treatment groups at 1-year post intervention adjusting for pre-intervention values and to estimate mean differences between treatment groups (95% CI). Medians and range (minimum, maximum values) will be used to describe non-normally distributed continuous data, Wilcoxon rank sum test will be used to compare treatment groups and Student t test to estimate mean differences (95% CI). Paired t tests will be used for differences between pre- and post-measurements. All analyses will be undertaken using SPSS version 24.0; and 0.05 defined statistical significance for all tests. Data will be analyzed on an intention- to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic stage 2 or greater (point C -1 or more pelvic organ prolapse quantification POP-Q) apical prolapse (uterovaginal or vault prolapse)
* Women with or without anterior compartment prolapse (point Ba -1 or more pelvic organ prolapse quantification POP-Q)
* Women without significant posterior compartment prolapse (point Bp -1 or more pelvic organ prolapse quantification POP-Q)

Exclusion Criteria:

* Women not eligible for surgery for medical or anesthesiological reasons
* Inability to comprehend questionnaires
* Inability to give informed consent
* Inability to return for review
* Prior laparoscopic prolapse repair
* Prior vaginal mesh prolapse procedure
* Vaginal length less than 6 cm.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Subjective cure rate of prolapse | at 12 months postoperatively
  Provided by the patient's feeling of the "Absence of a bulge in the vagina"
Objective success | at 12 months postoperatively
  Defined as anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total

SECONDARY OUTCOMES:
Patient global satisfaction | 1, 6, 12, 24 and 60 months
  This will be assessed using a Visual Analogue Scale for Global Satisfaction (10=very satisfies, 0=entirely dissatisfied)
Prolapse-related Quality of life | 1, 6, 12, 24 and 60 months
  This will be assessed using a validated questionnaire (Prolapse Quality of Life questionnaire P-QoL) The questionnaire contains 9 domains. Each answer of the patient will have values that range between 1 to 4 or 1 to 5 for the 1st question only). (1 very good 4/5 very poor). There is no overall score. A symptomatic woman might have only one domain impaired and another one might have all domains impaired. We consider both of them symptomatic but in different or same aspects of quality of life. To differentiate different domains, it is important for the decision of our surgery (we will be careful in shortening and narrowing a vagina of a woman who had only a preoperative high (impaired) Personal relationships domain score and other domains in the normal range).
  This will also help us in the follow up visits.
Perioperative complications | perioperatively
  This will be assessed using the Clavien-Dindo Scale. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life.
Sexual function | 1, 6, 12, 24 and 60 months
  This will be assessed using a validated questionnaire (Prolapse/Incontinence Sexual Questionnaire-IUGA revised PISQ-IR) The PISQ-IR is a validated evaluation tool which can be used clinically as well as in research for assessment of female sexual function (FSF), in women with female pelvic floor disorders. The resultant scale is composed of six sub-scales in sexually active (SA) women and four in women who are not sexually active (NSA).
  For women who are SA, it contains 21 items covering six domains: arousal/orgasm, partner related, condition specific, global quality rating, condition impact, and desire. For women who are not SA, it contains 12 items covering four domains: condition specific, partner related, global quality, and condition impact. Each domain receives a separate score
Patient satisfaction related to improvement of condition | 1, 6, 12, 24 and 60 months
  This will be assessed using the Patient Global Impression Scale of Improvement (PGI-I) (6=very much improved condition, 1=condition worsened)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barber MD, Maher C. Epidemiology and outcome assessment of pelvic organ prolapse. Int Urogynecol J. 2013 Nov;24(11):1783-90. doi: 10.1007/s00192-013-2169-9. PMID 24142054
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Handa VL, Garrett E, Hendrix S, Gold E, Robbins J. Progression and remission of pelvic organ prolapse: a longitudinal study of menopausal women. Am J Obstet Gynecol. 2004 Jan;190(1):27-32. doi: 10.1016/j.ajog.2003.07.017. PMID 14749630
- [Background] Morrill M, Lukacz ES, Lawrence JM, Nager CW, Contreras R, Luber KM. Seeking healthcare for pelvic floor disorders: a population-based study. Am J Obstet Gynecol. 2007 Jul;197(1):86.e1-6. doi: 10.1016/j.ajog.2007.02.051. PMID 17618770
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2016 Oct 1;10(10):CD012376. doi: 10.1002/14651858.CD012376. PMID 27696355
- [Background] Barber MD, Maher C. Apical prolapse. Int Urogynecol J. 2013 Nov;24(11):1815-33. doi: 10.1007/s00192-013-2172-1. PMID 24142057
- [Background] Vieillefosse S, Thubert T, Dache A, Hermieu JF, Deffieux X. Satisfaction, quality of life and lumbar pain following laparoscopic sacrocolpopexy: suture vs. tackers. Eur J Obstet Gynecol Reprod Biol. 2015 Apr;187:51-6. doi: 10.1016/j.ejogrb.2015.02.014. Epub 2015 Feb 18. PMID 25748488
- [Background] Dubuisson JB, Yaron M, Wenger JM, Jacob S. Treatment of genital prolapse by laparoscopic lateral suspension using mesh: a series of 73 patients. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):49-55. doi: 10.1016/j.jmig.2007.11.003. PMID 18262144
- [Background] Veit-Rubin N, Dubuisson JB, Gayet-Ageron A, Lange S, Eperon I, Dubuisson J. Patient satisfaction after laparoscopic lateral suspension with mesh for pelvic organ prolapse: outcome report of a continuous series of 417 patients. Int Urogynecol J. 2017 Nov;28(11):1685-1693. doi: 10.1007/s00192-017-3327-2. Epub 2017 Apr 17. PMID 28417156
- [Background] Digesu GA, Khullar V, Cardozo L, Robinson D, Salvatore S. P-QOL: a validated questionnaire to assess the symptoms and quality of life of women with urogenital prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2005 May-Jun;16(3):176-81; discussion 181. doi: 10.1007/s00192-004-1225-x. Epub 2004 Oct 21. PMID 15875234
- [Background] Veit-Rubin N, Digesu A, Swift S, Khullar V, Kaelin Gambirasio I, Dallenbach P, Boulvain M. Validation of the French version of the P-QoL questionnaire. Eur J Obstet Gynecol Reprod Biol. 2015 Sep;192:10-6. doi: 10.1016/j.ejogrb.2015.05.028. Epub 2015 Jun 10. PMID 26142910
- [Background] Digesu GA, Santamato S, Khullar V, Santillo V, Digesu A, Cormio G, Loverro G, Selvaggi L. Validation of an Italian version of the prolapse quality of life questionnaire. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):184-92. doi: 10.1016/s0301-2115(02)00229-4. PMID 12551790